CLINICAL TRIAL: NCT06511076
Title: An Open-Label, Single Center, Randomized, 2-Way Crossover, Single-Dose, Bioequivalence Study of Zilucoplan Injected Subcutaneously Either by a Prefilled Syringe or an Auto-Injector in Healthy Adult Participants
Brief Title: A Study to Evaluate Zilucoplan Injected Subcutaneously Either by a Prefilled Syringe or an Auto-injector in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DV0012
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers
MeSH Terms: interventions — zilucoplan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence AB (Experimental): Study participants randomized to this arm will receive a single subcutaneous (sc) injection of zilucoplan using pre-filled syringe (ZLP-PFS; Treatment A) as reference and a single sc injection of zilucoplan using an autoinjector (ZLP-AI; Treatment B) as test in the treatment sequence A-B on Day 1 of each Treatment Period.
  Interventions: Drug: Zilucoplan
- Treatment Sequence BA (Experimental): Study participants randomized to this arm will receive a single sc injection of zilucoplan using pre-filled syringe (ZLP-PFS; Treatment A) as reference and a single sc injection of zilucoplan using an autoinjector (ZLP-AI; Treatment B) as test in the treatment sequence B-A on Day 1 of each Treatment Period.
  Interventions: Drug: Zilucoplan

INTERVENTIONS:
Drug: Zilucoplan — Participants will receive a single sc injection of zilucoplan in the pre-specified sequence.
  Other Names: RA101495

SUMMARY:
The purpose of this study is to assess the bioequivalence pharmacokinetics, safety, tolerability and device deficiencies of zilucoplan (ZLP) in healthy adult participants

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Participants must be vaccinated with a quadrivalent vaccine and serogroup B vaccine against meningococcal infections (N. meningitidis) at least 2 weeks before the first administration of IMP if not previously vaccinated within 3 years prior to the start of IMP administration. Study participants who are not previously vaccinated may receive Menactra® (quadrivalent vaccine) and Bexsero® (serogroup B vaccine) during the Screening Period, 2 weeks prior to initiating IMP.
* Body mass index (BMI) ≥18.5 to ≤30.0kg/m2 at the Screening Visit.
* Male and/or female:
* A male participant must agree to use contraception during the Treatment Period as detailed in Appendix 4 of the protocol and for at least 40 days (approximately 5 half lives) after the last dose of IMP and refrain from donating sperm during this period.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:
* Not a female/woman of childbearing potential (WOCBP) OR
* A WOCBP who agrees to follow the contraceptive guidance during the Treatment Period and for at least 40 days (approximately 5 half lives), corresponding to time needed to eliminate IMP after the last dose of IMP.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form and in the protocol.

Exclusion Criteria:

* Participant has a history of or current significant medical disorder, psychiatric disorder, or laboratory abnormality that in the opinion of the Investigator makes the study participant unsuitable for participation in the study, including any previous or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking IMP; or interfering with the interpretation of data.
* Current or recent systemic infection within 2 weeks before the first administration of IMP or infection requiring intravenous antibiotics within 4 weeks before the first administration of IMP.
* Current history of alcohol or drug use disorder, as defined in Diagnostic and Statistical Manual of Mental Disorders V, within the previous 6 months.
* Participant has a known hypersensitivity to any components of the IMP or comparative drugs (and/or an investigational device) as stated in the protocol.
* Intended use of over-the-counter or prescription medication, vitamins, herbal/traditional medicines (including St John's Wort) or dietary supplements (excluding medicines for external use), with the exception of those specified in the Protocol, within 2 weeks before the first administration of IMP.
* Participant has used hepatic enzyme-inducing drugs (eg, glucocorticoids, phenobarbital, isoniazid, phenytoin, rifampicin) within 2 months before the first administration of IMP.
* Participant has previously participated in this study or participant has previously been assigned to treatment in a study of the medication under investigation in this study.
* Participant has participated in another study of an IMP (and/or an investigational device) within the previous 30 days or 5 half-lives (whichever is longer), or is currently participating in another study of an IMP (and/or an investigational device).
* Participants with clinically relevant abnormalities in a standard 12-lead electrocardiogram (ECG) at the Screening Visit as judged by the Investigator.
* Presence of hepatitis B surface antigen at the Screening Visit or within 3 months prior to dosing.
* Positive hepatitis C antibody test result at the Screening Visit or within 3 months prior to starting IMP. NOTE: Participants with positive hepatitis C antibody due to prior resolved disease can be enrolled if a confirmatory negative hepatitis C ribonucleic acid (RNA) test is obtained.
* Positive hepatitis C RNA test result at the Screening Visit or within 3 months prior to first dose of IMP. NOTE: Test is optional and participants with negative hepatitis C antibody test are not required to also undergo hepatitis C RNA testing.
* Positive human immunodeficiency virus antibody test at the Screening Visit.
* Positive syphilis test at the Screening Visit.
* Positive throat swab for N. meningitidis at the Screening Visit or a prior history of meningitis.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (1):
- DV0012 1, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, individual patient-level data cannot be adequately anonymized as there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in August 2024 and concluded in November 2024.
Pre-assignment Details: The Participant Flow refers to the All randomized Study Participants.
Groups:
- Sequence: Treatment A (ZLP-PFS) - Treatment B (ZLP-AI): Participants received a single subcutaneous (sc) injection in abdomen using zilucoplan pre-filled syringe (ZLP-PFS) (Treatment A) on Day 1 of Period 1 and a single sc injection in abdomen using zilucoplan auto-injector (ZLP-AI) (Treatment B) on Day 1 of Period 2 in the treatment sequence A-B. Each treatment period was of 35 days and was separated by 7-Days Washout period.
- Sequence: Treatment B (ZLP-AI) - Treatment A (ZLP-PFS): Participants received a single sc injection using ZLP-AI (Treatment B) on Day 1 of Period 1 and a single sc injection in abdomen using ZLP-PFS (Treatment A) on Day 1 of Period 2 in the treatment sequence B-A. Each treatment period was of 35 days and was separated by 7-Days Washout period.
Period: Treatment Period 1 (35 Days)
Arm/Group | Sequence: Treatment A (ZLP-PFS) - Treatment B (ZLP-AI) | Sequence: Treatment B (ZLP-AI) - Treatment A (ZLP-PFS)
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Treatment Period 2 (35 Days)
Arm/Group | Sequence: Treatment A (ZLP-PFS) - Treatment B (ZLP-AI) | Sequence: Treatment B (ZLP-AI) - Treatment A (ZLP-PFS)
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline refers All Randomized Study Participants which consisted of all study participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence: Treatment A (ZLP-PFS) - Treatment B (ZLP-AI) | Sequence: Treatment B (ZLP-AI) - Treatment A (ZLP-PFS) | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.0 (5.9) | 36.1 (15.9) | 30.8 (10.0)
Age, Customized [Count of Participants; unit: Participants]
  18 - <65 years | 7 | 7 | 14
  65 - <85 years | 0 | 0 | 0
  >=85 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 3 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  White | 5 | 7 | 12
  Other or Mixed | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero (Predose [Day 1]) to Infinity (AUC) for Zilucoplan
Description: AUC was defined as the area under the plasma concentration-time curve from time zero (predose [Day 1]) to infinity for zilucoplan.
Time Frame: Baseline (Day 1 of each treatment period at predose) and at predefined time points up to 816 hours (Day 35) postdose
Population: The Pharmacokinetic (PK) Set consisted of all study participants who were randomized, received at least 1 dose of ZLP, and had at least 1 observable PK concentration measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliters (h*ng/mL)
Groups:
- ZLP-PFS: Participants received a single sc injection of zilucoplan using pre-filled syringe (ZLP-PFS; Treatment A) on Day 1 of Treatment Period 1 and 2.
- ZLP-AI: Participants received a single sc injection using ZLP-AI (Treatment B) on Day 1 of Treatment Period 1 and 2.
Arm/Group | ZLP-PFS | ZLP-AI
Number analyzed (Participants) | 14 | 14
hour*nanogram per milliliters (h*ng/mL) | 950930 (15.0) | 932740 (17.1)
Statistical Analysis 1: Comparison: ZLP-PFS vs ZLP-AI; Test type: Equivalence — Bioequivalence was concluded if the 90% CIs for the ratio of the geometric means of Treatment ZLP-AI (test [T]) / Treatment ZLP-PFS (Reference [R]) were included in the range from 0.80 - 1.25; Mixed Effects model; GLSM ratio = 0.9809, 90% CI [0.9529 to 1.0097] — The GLSM ratio was calculated: ZLP-AI/ZLP-PFS

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 (Predose [Day 1]) to the Time of the Last Quantifiable Concentration (AUC[0-t]) for Zilucoplan
Description: AUC(0-t) was defined as the area under the plasma concentration-time curve from time 0 (predose [Day 1]) to the time of the last quantifiable concentration for zilucoplan.
Time Frame: Baseline (Day 1 of each treatment period at predose) and at predefined time points up to 816 hours (Day 35) postdose
Population: The PK Set consisted of all study participants who were randomized, received at least 1 dose of ZLP, and had at least 1 observable PK concentration measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | ZLP-PFS | ZLP-AI
Number analyzed (Participants) | 14 | 14
h*ng/mL | 921190 (14.5) | 904500 (16.4)
Statistical Analysis 1: Comparison: ZLP-PFS vs ZLP-AI; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Effects model; GLSM Ratio = 0.9819, 90% CI 2-sided [0.9543 to 1.0102] — The GLSM ratio was calculated: ZLP-AI/ZLP-PFS

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for Zilucoplan
Description: Cmax was defined as the maximum observed plasma concentration for zilucoplan.
Time Frame: Baseline (Day 1 of each treatment period at predose) and at predefined time points up to 816 hours (Day 35) postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliters (ng/mL)
Arm/Group | ZLP-PFS | ZLP-AI
Number analyzed (Participants) | 14 | 14
nanograms per milliliters (ng/mL) | 5599.8 (11.3) | 5597.6 (11.0)
Statistical Analysis 1: Comparison: ZLP-PFS vs ZLP-AI; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Effects model; GLSM ratio = 0.9996, 90% CI 2-sided [0.9594 to 1.0416] — The GLSM ratio was calculated: ZLP-AI/ZLP-PFS

4. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) From Day 1 up to the End of Study (EOS) Visit or Early Termination (ET) Visit
Description: An AE was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of investigational medicinal product, whether or not considered related to the investigational medicinal product. A TEAE was defined as any AE with a start date/time on or after the administration of IMP in each Treatment Period, and up to and including 40 days after the single dose in each Treatment Period (or up to the first dose in Period 2 (for TEAEs following the first dose in Period 1) or last contact date (for TEAEs following the first dose in Period 2) depending on which occurs first. Percentages were displayed to one decimal place and was correspond to whole participant counts due to rounding.
Time Frame: From Day 1 to EOS visit or ET visit (up to 82 days)
Population: The safety set (SS) consisted of all study participants who were randomized and receive at least 1 dose of ZLP. Study participants were classified according to the sequence to which they were randomly assigned.
Measure: Number; unit: percentage of participants
Arm/Group | ZLP-PFS | ZLP-AI
Number analyzed (Participants) | 14 | 14
percentage of participants | 57.1 | 57.1

5. Secondary Outcome: Percentage of Participants With Serious Treatment-emergent Adverse Events (Serious TEAEs) From Day 1 up to the End of Study (EOS) Visit or Early Termination (ET) Visit
Description: An SAE was defined as any untoward medical occurrence that, at any dose, met 1 or more of the criteria listed:
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Is a congenital anomaly/birth defect
  * Important medical events such as (but not limited to) invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias, convulsions not resulting in hospitalization, or development of intervention dependency or intervention abuse.
Time Frame: From Day 1 to EOS visit or ET visit (up to 82 days)
Population: The SS consisted of all study participants who were randomized and receive at least 1 dose of ZLP. Study participants were classified according to the sequence to which they were randomly assigned.
Measure: Number; unit: percentage of participants
Arm/Group | ZLP-PFS | ZLP-AI
Number analyzed (Participants) | 14 | 14
percentage of participants | 0 | 0

6. Secondary Outcome: Percentage of Participants With Serious Adverse Device Effects (SADE) From Day 1 up to the End of Study (EOS) Visit or Early Termination (ET) Visit
Description: An SAE was defined as any untoward medical occurrence that, at any dose, met 1 or more of the criteria listed:
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Is a congenital anomaly/birth defect
  * Important medical events such as (but not limited to) invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias, convulsions not resulting in hospitalization, or development of intervention dependency or intervention abuse.
  A SADE was defined as an adverse device effect that has resulted in any of the consequences characteristic of a SAE.
Time Frame: From Day 1 to EOS visit or ET visit (up to 82 days)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | ZLP-PFS | ZLP-AI
Number analyzed (Participants) | 14 | 14
percentage of participants | 0 | 0

7. Secondary Outcome: Percentage of Participants With Non-serious Adverse Device Effects (ADE) From Day 1 up to the End of Study (EOS) Visit or Early Termination (ET) Visit
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory finding) in study participants, users, or other persons, whether or not related to the investigational medical device. An ADE was defined as an AE related to the use of an investigational medical device.
Time Frame: From Day 1 to EOS visit or ET visit (up to 82 days)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | ZLP-PFS | ZLP-AI
Number analyzed (Participants) | 14 | 14
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 to EOS visit or ET visit (up to 82 days)
Description: A TEAE was defined as any AE with a start date/time on or after the administration of IMP in each Treatment Period, and up to and including 40 days after the single dose in each Treatment Period (or up to the first dose in Period 2 (for TEAEs following the first dose in Period 1) or last contact date (for TEAEs following the first dose in Period 2) depending on which occurs first.
Arm/Group | ZLP-PFS | ZLP-AI
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 8/14 | 8/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZLP-PFS (N=14) | ZLP-AI (N=14)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 1 (1)
Catheter site papule (General disorders) | 1 (1) | 0 (0)
Catheter site pruritus (General disorders) | 1 (1) | 0 (0)
Catheter site related reaction (General disorders) | 1 (1) | 0 (0)
Catheter site swelling (General disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 5 (5)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nitrite urine present (Investigations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT06511076/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT06511076/SAP_001.pdf